CLINICAL TRIAL: NCT04807751
Title: A Phase 1 Clinical Trial to Evaluate the Photoallergic Potential of Delgocitinib Cream 20 mg/g After Topical Occlusive Application in Subjects With Healthy Skin
Brief Title: Clinical Trial to Evaluate UV-light-induced Allergic Skin Reactions After Application of Delgocitinib Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: LP0133-1411; 2020-003090-22 (EudraCT Number)
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: All subjects will receive all treatments with treatments randomised over test fields.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delgocitinib cream 20 mg/g (Experimental): topical occlusive administration
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream vehicle (Placebo Comparator): topical occlusive administration
  Interventions: Drug: Delgocitinib cream vehicle
- Untreated skin (No Intervention): topical occlusive administration

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application
  Other Names: LEO 124249 cream
  Arms: Delgocitinib cream 20 mg/g
Drug: Delgocitinib cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
  Arms: Delgocitinib cream vehicle

SUMMARY:
Participants will have study medicine applied by site staff- delgocitinib cream or vehicle, and then exposed to UV light. The trial is designed to find out if delgocitinib cream can cause skin photoallergy after UV-light exposure in people with healthy skin.

DETAILED DESCRIPTION:
This is a single-centre, randomised, double-blind, vehicle-controlled, within-subject comparison phase 1 trial in Germany.

The trial consists of a screening phase, an induction phase, a rest phase, and a challenge phase. There will be 2 columns of test fields on each participant's back with the 3 treatments in either column for a total of 6 treatments. One column of test fields will be irradiated and the other will not be irradiated. All participants will be exposed to UV-light on skin treated delgocitinib cream or vehicle and on untreated skin on test fields to be irradiated.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy subjects aged 18-64 years (inclusive).
* Fitzpatrick skin type of I, II, or III.

Exclusion Criteria:

* Atopic dermatitis, eczema, psoriasis, acne, dermatitis solaris or suntan that could interfere with the test field evaluation, hyperpigmentation, multiple naevi, tattoos, blemishes, or dense body hair in the range of the test fields.
* Any other skin disease or other visible skin condition noted on physical examination which in the investigator's opinion might interfere with the evaluation of the test field reaction.
* Any history of or presence of cancerous or precancerous skin lesions in general including melanoma, lentigo maligna, basal cell carcinoma, dysplastic naevi or actinic keratoses.
* History of or active or both photo-induced or photo-aggravated disease (e.g. cutaneous or lupus erythematodes, polymorphic light eruptions).
* Use of any topical or systemic medication that could interfere with the trial objective within 2 weeks before randomisation until subject's end of trial.
* Use of drugs that might cause photosensitising or phototoxic reactions within 4 weeks before randomisation until subject's end of trial.
* Foreseeable intensive UV-light exposure to test fields within 4 weeks before randomisation until subject's end of trial (solar or artificial).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Positive skin reaction at 72 hours after irradiation | Up to 72 hours after irradiation
  A reaction is considered positive if the skin reaction score for the irradiated test field is at least 1 point higher than both the non-irradiated test field exposed to the same strength of IMP, and the irradiated control field.
  The evaluation of skin reaction at the end of the challenge phase performed using the following scale:
  * 0 negative
  * 1 equivocal
  * 2 positive. A positive score indicates presence of a UV-light-induced allergic skin reaction.

SECONDARY OUTCOMES:
Number of adverse events from baseline to 14 days after subject's end of trial | From baseline to 14 days after subject's end of trial (Day 5 of challenge phase, or if applicable Day 5 of re-challenge phase.
  Treatment-emergent adverse event
Skin reaction score after irradiation during induction phase | up to Day 22
  A reaction is considered positive if the skin reaction score for the irradiated test field is at least 1 point higher than both the non-irradiated test field exposed to the same strength of IMP, and the irradiated control field.
  The grading for the skin reaction score will be performed according to the following 5-point scale:
  * 0 No reaction
  * 1 Erythema
  * 2 Erythema with dermal infiltrate
  * 3 Erythema with papulovesicles
  * 4 Erythema with blisters, erosions
Skin reaction score after irradiation during the challenge phase (up to Day 40, Week 6). | up to Day 40
  A reaction is considered positive if the skin reaction score for the irradiated test field is at least 1 point higher than both the non-irradiated test field exposed to the same strength of IMP, and the irradiated control field.
  The grading for the skin reaction score will be performed according to the following 5-point scale:
  * 0 No reaction
  * 1 Erythema
  * 2 Erythema with dermal infiltrate
  * 3 Erythema with papulovesicles
  * 4 Erythema with blisters, erosions

CONTACTS AND LOCATIONS:
Locations (1):
- Bioskin Research Center Dermatology, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No